CLINICAL TRIAL: NCT02719990
Title: An Open-Label, Long-Term Extension Study of the Safety of Somavaratan (VRS-317) in Adults With Growth Hormone Deficiency (GHD)
Brief Title: Open-label Extension Study to Evaluate the Safety of Long-term Twice-monthly Administration of Somavaratan in Adult Growth Hormone Deficiency (AGHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Phase 3 clinical trial of somavaratan in pediatric growth hormone deficiency (PGHD) did not meet its primary endpoint of non-inferiority.
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Organization: Aravive, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15VR8
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Adult Growth Hormone Deficiency (AGHD)
Keywords: VRS-317; Long Acting Growth Hormone; Versartis; somavaratan; Growth Hormone Deficiency; Adult Growth Hormone Deficiency; AGHD; Growth Hormone Replacement; Growth Hormone Replacement Therapy; XTEN
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somavaratan (Experimental): Long-acting recombinant human growth hormone therapy administered subcutaneously twice-monthly in adult participants with GHD
  Interventions: Drug: somavaratan

INTERVENTIONS:
Drug: somavaratan — Long-acting recombinant human growth hormone therapy administered subcutaneously twice-monthly
  Other Names: VRS-317

SUMMARY:
Open-label extension study to evaluate the safety of long-term twice-monthly administration of somavaratan in adults with Growth Hormone Deficiency (GHD).

DETAILED DESCRIPTION:
An open-label extension study to evaluate the safety of long-term twice-monthly administration of somavaratan in adults with GHD. This multicenter study is open to participants completing a Versartis adult GHD study as well as approximately 40 new somavaratan naïve participants (either recombinant human growth hormone [rhGH] treatment naïve or currently receiving daily rhGH therapy). All participants will receive twice-monthly (every 15 days ± 2 days) subcutaneous (SC) somavaratan. Doses will be titrated to each participant's individual insulin-like growth factor-I (IGF-I) responses based on the IGF-I level 7 days post-dose until a maintenance dose is achieved. Participants receiving somavaratan in a previous somavaratan study will have their dose decreased by half (minimum dose of 20 milligrams [mg], 40 mg for women on estrogen, rounded down to the nearest even number) and will be titrated per the Dose Titration Plan. New participants enrolling in this study will be assigned to one of two cohorts based on sensitivity to rhGH and titrated per the Dose Titration Plan.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of childbearing potential must have negative pregnancy test and use appropriate contraceptive methods
* Documented GHD during adulthood
* Participants naive to somavaratan must have an IGF-1 SDS value ≤ 0 at Screening
* Participants taking other hormone replacement therapy must have been on a stable course of treatment for at least 3 months
* Underlying disorders responsible for the participant's GHD must have been clinically stable for at least 6 months
* Participants receiving daily rhGH injections must washout for ≥ 14 days
* Body mass index (BMI) (kilograms [kg]/meter square [m^2]) between 18.0 and 40.0

Exclusion Criteria:

* Untreated adrenal insufficiency
* Recently diagnosed thyroid dysfunction which is not being treated or has not been stable on therapy for at least 3 months
* Currently taking anti-inflammatory dose of glucocorticoids that could potentially compromise safety or efficacy assessments
* Currently taking a GHRH or IGF-I product
* Current significant cardiovascular disease, heart insufficiency of New York Heart Association (NYHA) class > 2
* Current significant disease thought to increase risk of receiving growth hormone or confound assessment of study outcomes
* History of diabetes mellitus or inadequate glucose control
* Current drug or alcohol abuse
* Current human immunodeficiency virus (HIV) wasting syndrome (HIV testing not required)
* History of malignancy in adulthood (participants with a history of childhood malignancy that were subsequently treated with rhGH in childhood and remain GHD in adulthood may be enrolled)
* Women who are pregnant or breastfeeding
* Treatment with an investigational drug other than somavaratan within 30 days prior to Screening
* A significant abnormality in Screening laboratory results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Sponsor GmbH

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was open to participants completing a Versartis adult growth hormone deficiency (GHD) study (15VR7 [NCT02526420]) as well as new somavaratan naïve participants (either recombinant human growth hormone [rhGH] treatment naïve or receiving daily rhGH therapy).
Groups:
- Somavaratan: Participants received once-monthly subcutaneous (SC) somavaratan per Protocol Version 1.0. The dosing regimen was then modified in Protocol Version 2.0 to twice-monthly SC somavaratan. Doses were titrated to each participant's individual IGF-I responses based on the insulin-like growth factor-I (IGF-I) level 7 days postdose until a maintenance dose was achieved. Maintenance dose was defined as an IGF-I value between 0 and 2.0 standard deviation score (SDS) for two consecutive 7-day postdose time points (Day 8, peak level). Participants who received somavaratan once-monthly in this study or in a previous somavaratan study (15VR7), had their dose decreased by half (minimum dose of 20 milligrams [mg], 40 mg for women on estrogen, rounded down to the nearest even number) and were titrated based on IGF-I level at Day 8. New participants enrolling in this study received a starting dose of 20 mg twice-monthly (40 mg for women on estrogen) and were titrated based on IGF-I level at Day 8. Maintenance doses were adjusted further based on pharmacodynamic (PD) data at the discretion of the Investigator or Medical Monitor. The maximum allowable dose of somavaratan was 250.0 mg.
Period: Overall Study
Arm/Group | Somavaratan
Started | 36
Received at Least 1 Dose of Study Drug | 36
Completed | 0
Not Completed | 36
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Study Terminated By Sponsor | 32

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of study drug.
Groups:
- Somavaratan: Participants received once-monthly SC somavaratan per Protocol Version 1.0. The dosing regimen was then modified in Protocol Version 2.0 to twice-monthly SC somavaratan. Doses were titrated to each participant's individual IGF-I responses based on the IGF-I level 7 days postdose until a maintenance dose was achieved. Maintenance dose was defined as an IGF-I value between 0 and 2.0 SDS for two consecutive 7-day postdose time points (Day 8, peak level). Participants who received somavaratan once-monthly in this study or in a previous somavaratan study (15VR7), had their dose decreased by half (minimum dose of 20 mg, 40 mg for women on estrogen, rounded down to the nearest even number) and were titrated based on IGF-I level at Day 8. New participants enrolling in this study received a starting dose of 20 mg twice-monthly (40 mg for women on estrogen) and were titrated based on IGF-I level at Day 8. Maintenance doses were adjusted further based on PD data at the discretion of the Investigator or Medical Monitor. The maximum allowable dose of somavaratan was 250.0 mg.
Arm/Group | Somavaratan
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: From first dose of study drug up to approximately 2 years
Population: Safety population included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Somavaratan
Number analyzed (Participants) | 36
Participants | 30

2. Secondary Outcome: Average Dose Level During Titration/Maintenance
Description: Total average dose received by a participant during titration/maintenance has been reported.
Time Frame: Up to Month 12
Population: Safety population included all participants who received any amount of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Somavaratan
Number analyzed (Participants) | 33
mg | 41.60 (47.398)

3. Secondary Outcome: Number of Participants With Dose Adjustments
Description: The number of participants with a dose adjustment (titrated up/down) at each month are summarized.
Time Frame: Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: Safety population included all participants who received any amount of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants analyzed at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Somavaratan
Number analyzed (Participants) | 11
Participants
  Month 2: Titrated Up | 11
  Month 2: Titrated Down | 0
  Month 3: number analyzed (Participants) | 7
  Month 3: Titrated Up | 7
  Month 3: Titrated Down | 0
  Month 4: number analyzed (Participants) | 8
  Month 4: Titrated Up | 6
  Month 4: Titrated Down | 2
  Month 5: number analyzed (Participants) | 5
  Month 5: Titrated Up | 3
  Month 5: Titrated Down | 2
  Month 6: number analyzed (Participants) | 3
  Month 6: Titrated Up | 3
  Month 6: Titrated Down | 0
  Month 7: number analyzed (Participants) | 3
  Month 7: Titrated Up | 3
  Month 7: Titrated Down | 0
  Month 8: number analyzed (Participants) | 4
  Month 8: Titrated Up | 3
  Month 8: Titrated Down | 1
  Month 9: number analyzed (Participants) | 0
  Month 9: Titrated Up | 0
  Month 9: Titrated Down | 0
  Month 10: number analyzed (Participants) | 0
  Month 10: Titrated Up | 0
  Month 10: Titrated Down | 0
  Month 11: number analyzed (Participants) | 3
  Month 11: Titrated Up | 1
  Month 11: Titrated Down | 2
  Month 12: number analyzed (Participants) | 1
  Month 12: Titrated Up | 0
  Month 12: Titrated Down | 1

4. Secondary Outcome: Number of Participants Who Were Anti-drug Antibody (ADA) Positive
Time Frame: Up to approximately 2 years
Population: Safety population included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Somavaratan
Number analyzed (Participants) | 36
Participants | 22

5. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies (NABs)
Time Frame: Up to approximately 2 years
Population: Safety population included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Somavaratan
Number analyzed (Participants) | 36
Participants | 15

6. Secondary Outcome: Change From Baseline in Mean Insulin-like Growth Factor 1 (IGF-I) Standard Deviation Score (SDS) at Specified Timepoints During Maintenance Period
Description: Changes in the IGF-I levels were assessed as Standard Deviation Scores (SDS). The SDS was calculated as the actual value of IGF-I minus mean reference value of IGF-1 divided by reference standard deviation of IGF-I. The mean and the standard deviation (SD) vary depending on the age and sex of the participant. Change in IGF-I level (SDS) at specified timepoints from baseline was assessed. A higher score reflects a better outcome.
Time Frame: Baseline, Month 2 Day 1, Month 2 Day 8, Month 3 Day 1, Month 3 Day 8, Month 4 Day 1, Month 4 Day 8, Month 5 Day 1, Month 5 Day 8, Month 6 Day 1, Month 6 Day 8, Month 7 Day 1, Month 7 Day 8, Month 8 Day 1, Month 8 Day 8, Month 10 Day 1, and Month 10 Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Somavaratan
Number analyzed (Participants) | 18
SDS
  Month 2 Day 1: number analyzed (Participants) | 15
  Month 2 Day 1 | 0.76 (0.639)
  Month 2 Day 8: number analyzed (Participants) | 16
  Month 2 Day 8 | 1.83 (0.899)
  Month 3 Day 1: number analyzed (Participants) | 14
  Month 3 Day 1 | 0.45 (0.457)
  Month 3 Day 8: number analyzed (Participants) | 14
  Month 3 Day 8 | 1.44 (0.915)
  Month 4 Day 1 | 0.49 (0.751)
  Month 4 Day 8 | 1.73 (1.221)
  Month 5 Day 1: number analyzed (Participants) | 3
  Month 5 Day 1 | 0.18 (0.738)
  Month 5 Day 8: number analyzed (Participants) | 4
  Month 5 Day 8 | 1.68 (0.691)
  Month 6 Day 1: number analyzed (Participants) | 3
  Month 6 Day 1 | 0.74 (0.500)
  Month 6 Day 8: number analyzed (Participants) | 3
  Month 6 Day 8 | 1.38 (0.777)
  Month 7 Day 1: number analyzed (Participants) | 13
  Month 7 Day 1 | 0.74 (0.541)
  Month 7 Day 8: number analyzed (Participants) | 12
  Month 7 Day 8 | 1.82 (1.414)
  Month 8 Day 1: number analyzed (Participants) | 1
  Month 8 Day 1 | 0.30
  Month 8 Day 8: number analyzed (Participants) | 1
  Month 8 Day 8 | 4.30
  Month 10 Day 1: number analyzed (Participants) | 10
  Month 10 Day 1 | 0.91 (0.845)
  Month 10 Day 8: number analyzed (Participants) | 9
  Month 10 Day 8 | 1.76 (1.539)

7. Secondary Outcome: Mean Insulin-like Growth Factor-binding Protein 3 (IGFBP-3) SDS During Maintenance Period
Time Frame: Baseline up to Month 12
Population: Due to early termination of study, no data were collected for this outcome measure.
Arm/Group | Somavaratan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 2 years
Description: Safety population included all participants who received any amount of study drug.
Arm/Group | Somavaratan
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somavaratan (N=36)
Adrenal insufficiency (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somavaratan (N=36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Hernia (General disorders) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Pharyngitis (Infections and infestations) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Gastroenteritis (Infections and infestations) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Hordeolum (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 3
Fall (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Diverticulitis (Infections and infestations) | 2
Very low density lipoprotein increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 2
C-reactive protein increased (Investigations) | 3
Nasopharyngitis (Infections and infestations) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Sinusitis (Infections and infestations) | 2
Blood phosphorus decreased (Investigations) | 1
Blood phosphorus increased (Investigations) | 2
Nausea (Gastrointestinal disorders) | 3
Viral pharyngitis (Infections and infestations) | 1
Blood potassium decreased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Haemangioma removal (Surgical and medical procedures) | 1
Injection site erythema (General disorders) | 1
Fatigue (General disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Macule (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Gastroenteritis viral (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Influenza (Infections and infestations) | 1
White blood cell count increased (Investigations) | 1
Abdominal wall mass (Gastrointestinal disorders) | 1
Migraine (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Injection site reaction (General disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 2
Viral upper respiratory tract infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Oral candidiasis (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Oral herpes (Infections and infestations) | 1
Depression (Psychiatric disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Skin lesion excision (Surgical and medical procedures) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Oedema peripheral (General disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Choroidal detachment (Eye disorders) | 1
Stress (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Weight increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
US Sites:

Institution shall cause Principal Investigator to submit a complete copy of the proposed publication to Sponsor at least 60 days prior to presentation or submission to any third party.

Non-US sites:

The Investigator and the Institution agree that any proposed publication relating to the research and/or Study conducted under this Agreement will be submitted to Sponsor for review at least 90 days prior to submission for publication.

Additional agreement conditions apply.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02719990/Prot_SAP_000.pdf